CLINICAL TRIAL: NCT03487523
Title: Health Message Framing to Improve Uptake of Bowel Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Heatlh Service Ayrshire and Arran (Other Government)
Responsible Party: Principal Investigator, Patrick McGuire, GP Registrar, National Heatlh Service Ayrshire and Arran
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 224710
Record Dates: First submitted 2018-02-02; First posted 2018-04-04 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Colorectal Cancer
Keywords: Behavioural Economics
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be a cross sectional randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention 1 (Active Comparator): Text message (SMS Message)
  Interventions: Behavioral: Text Message
- Intervention 2 (Active Comparator): Text message (SMS Message)
  Interventions: Behavioral: Text Message
- Intervention 3 (No Intervention): no intervention

INTERVENTIONS:
Behavioral: Text Message — As already stated
  Arms: Intervention 1; Intervention 2

SUMMARY:
The objective of this research is to investigate whether a text message (SMS message) prompting participation in the UK national bowel cancer screening programme improves uptake for those who have not responded to the test.

The secondary objective is to investigate whether the framing/phrasing of the text message improves participation , whether by stating the benefits of uptake or alternatively by stating the costs of non-uptake.

DETAILED DESCRIPTION:
A national register exists for GP practices to identify which patients of theirs have or have not participated in a national bowel cancer screening programme. A sample of 1600 patients belonging to a particular practice in Scotland aged between 50 and 74 have been identified as having received the test kit but have not responded to it. These individuals have also previously consented to being contacted by the practice via phone text/SMS message for reminders.

The sample will be randomised into three equally populated groups:

* One group will act as the control arm and will receive no text message.
* One group will receive a text message which encourages participation in the screening programme and provides information on the cost of not participating (negative frame) - "If you do not take part in screening then you increase the risk of having an undiagnosed tumor."
* One group will receive a text message which encourages participation in the screening programme and provides information on the benefit of participating (positive frame) - "If you take part in screening then you decrease the risk of having an undiagnosed tumor."

Both text messages will include a weblink which will direct individuals receiving the text to find more information and also with instructions on how to order another kit should they have misplaced the kit that was mailed out to them.

The observation period will last 6 months and patients receiving the text will receive 3 texts in total. One at the start of the 6 months and another every two months after that. These messages will not change or alternate, that is the negatively framed group will receive the same text once every 2 months on 3 occasions in total and vice versa. Other studies have used shorter intervals between text messages to encourage change, although 6 months to 1 year is a standard amount of time overall. The researchers feel that while more regular messages may be more likely prompt behaviour there is also a risk of over-burdening the patient with reminders, as such 3 texts over 6 months was decided upon as a reasonable frequency.

At the end of the 6 months data on uptake of screening for those 1600 patients during that time will be extracted by the practice clinician, matched with patient characteristics (e,g, age, sex) and anonymised so that patients cannot be identified. This will then be sent to the health economist to analyse the data and test the hypotheses above. Regression analysis will be used to see whether a differential pattern of uptake exists between groups receiving and not receiving the text message.

Once analysed the results will be fed back to the practice in order to help inform future reminders and will also be drafted into a paper to be submitted for peer-review.

ELIGIBILITY:
Inclusion Criteria:

* Over 55
* Not yet returned a bowel cancer screening sample
* No diagnosis of bowel cancer

Exclusion Criteria:

* Under 55
* Have already completed bowel cancer screening
* Diagnosed with bowel cancer

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2018-06-21 (Estimated); Primary Completion 2018-12-21 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants taking part in the Scottish national bowel cancer screening programme | 6 months
  Number of participants taking part in the Scottish national bowel cancer screening programme represented as a patient having submitted a faecal occult blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGuire, Principal Investigator — Dr

IPD SHARING:
Plan to Share IPD: No